CLINICAL TRIAL: NCT00116480
Title: Misoprostol in the Treatment of Post Partum Hemorrhage: A Placebo Randomised Controlled Trial in 4 Karachi Hospitals
Brief Title: Misoprostol in the Treatment of Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Aga Khan University (Other); Aga Khan Health Services (Other); The Aga Khan Foundation (Other); Family Care International (Other)
Responsible Party: Gynuity Health Projects, Gynuity Health Projects
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2.4.2
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum Haemorrhage; Misoprostol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Experimental): three tablets of active misoprostol (600 mcg) given sublingually
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): three tablets resembling misoprostol given sublingually
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 600 mcg of sublingual misoprostol

SUMMARY:
Postpartum haemorrhage (PPH) remains a leading cause of maternal mortality, despite treatment with conventional methods. Uncontrolled reports and three small randomised controlled trials have suggested that misoprostol may have an additive effect to routine treatment, and there is a serious danger that this method will be used widely without research to document the effectiveness or risks of this method. In this randomised controlled trial (RCT), we propose to test whether 600 μg of sublingually administered misoprostol in women requiring additional uterotonics after delivery, and after routine syntocinon to all women during or after delivery, has additional effects above the additional conventional uterotonics in reducing PPH. Women with measured blood loss greater than or equal to 500 mls in 4 Karachi hospitals who give consent will be given locally routine treatment for PPH. In addition, they will be enrolled by drawing the next of a series of randomised treatment packs containing misoprostol or placebo. The primary outcome measure will be blood loss greater than or equal to 500 mls after enrolment.

ELIGIBILITY:
Inclusion Criteria:

* All women delivering vaginally with clinically diagnosed PPH requiring uterotonics

Exclusion Criteria:

* Refusal to give consent for participation or if the woman is too distressed to give consent
* Woman is not entitled to give informed consent (e.g. minors without a guardian)
* Woman who had a caesarean section
* Delivery is regarded as abortion (gestational age < 28 weeks)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-12; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Blood loss greater than or equal to 500 mls after enrolment | Blood loss measured for minimum of 1 hour or until active bleeding ceased

SECONDARY OUTCOMES:
Average blood loss | Blood loss measured for minimum of one hour or until active bleeding ceased
Clinical complications (need for transfusion, hysterectomy) | After delivery and prior to hospital discharge
Pre-delivery and post-delivery hemoglobin measures | Pre-delivery hemoglobin measured upon admission to hospital (during labor) and measured postpartum 12-24 hours after delivery
Side effects | observed or reported following study treatment and prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem F Zuberi, MD, Principal Investigator — Aga Khan University Hospital, Karachi
Locations (2):
- Pakistan (2):
  - Aga Khan University Hospital, Karachi
  - The Aga Khan Health Services, Karachi

REFERENCES:
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518
- [Derived] Zuberi NF, Durocher J, Sikander R, Baber N, Blum J, Walraven G. Misoprostol in addition to routine treatment of postpartum hemorrhage: a hospital-based randomized-controlled trial in Karachi, Pakistan. BMC Pregnancy Childbirth. 2008 Aug 21;8:40. doi: 10.1186/1471-2393-8-40. PMID 18718007
- See also: Related Info — http://www.gynuity.org